CLINICAL TRIAL: NCT06689423
Title: Clinical Performance Evaluation of the VitaSIRO Solo™ SARS-CoV-2/Flu/RSV Assay
Brief Title: Clinical Evaluation of the VitaSIRO Solo™ Respiratory Assay
Status: Not yet recruiting | Type: Observational
Sponsor: Credo Diagnostics Biomedical Pte. Ltd. (Industry)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: B-AO-11-011
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2; COVID-19; RSV; Influenza
Keywords: Respiratory; SARS-CoV-2; COVID-19; Influenza; RSV; POCT
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover nasal swab (NS) and nasopharyngeal swab (NPS) specimens will be frozen and shipped back to sponsor for storage which might be used for future assay development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptomatic Cohort: Subjects displaying signs and/or symptoms of respiratory tract infections
  Interventions: Device: Credo POCT Device

INTERVENTIONS:
Device: Credo POCT Device — Testing Credo's POCT device for respiratory viruses detection.

SUMMARY:
The purpose of this clinical trial is to demonstrate the clinical performance of the VitaSIRO solo™ SARS-CoV-2/Flu/RSV Assay in detecting SARS-CoV-2, Flu A, Flu B and RSV in symptomatic population. The primary aim is to determine the PPA/NPA against a comparator assay. The secondary aim is to determine the diagnostic sensitivity, specificity, PPV and NPV against the standard-of-care test. Each subjects will be asked to provide both nasal swab (NS) and nasopharyngeal swab (NPS) for testing purposes.

DETAILED DESCRIPTION:
The study is designed as a multisite, observational, prospective study. Subjects will be prospectively recruited from the target population, specifically individuals displaying signs and/or symptoms of respiratory tract infections. Consent for participation will be obtained prior to any eligibility confirmation or sample collection. Subsequently, both nasal swab (NS) and nasopharyngeal swab (NPS) specimens will be collected from each subject. These specimens will be tested using both the VitaSIRO solo™ SARS-CoV-2/Flu/RSV Assay and the Cepheid Xpert Xpress CoV-2/Flu/RSV plus assay (comparator) to determine the Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA).

Subjects will be recruited across up to 20 sites, targeting the following intended user groups:

Trained laboratory professionals in a central laboratory setting Trained healthcare practitioners in a point-of-care (POC) setting under CLIA moderate and high complexity.

If a standard-of-care (SOC) diagnosis is available, the sensitivity, specificity, Positive Predictive Value (PPV), and Negative Predictive Value (NPV) will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subject displaying one or more of the following signs and/or symptoms of a respiratory tract infection:

  1. Fever
  2. Cough
  3. Nasal Congestion
  4. Shortness of breath
  5. Difficulty in breathing
  6. Runny nose
  7. Sore throat
  8. Muscle pain
  9. Headache
  10. Chills
  11. Nausea
  12. Diarrhoea
  13. Vomiting
  14. New loss of taste/smell
* If age 18 or over, subject is willing and capable of providing written informed consent. If under the age of 18, parent or legal guardian is willing to and capable of providing consent/assent. Assent should be obtained from minor subjects of appropriate intellectual age as defined by the IRB.

Exclusion Criteria:

* Subject is unable to provide consent and assent (as appropriate) or parental/legal guardian consent permission and assent (as appropriate) cannot be obtained.
* PI determines that specimen collection represents an unacceptable risk.
* Subjects who have already been enrolled in the study previously.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects involved in the study include individuals displaying signs and/or symptoms of respiratory tract infections as per the intended purpose of the VitaSIRO solo™ SARS-CoV-2/Flu/RSV Assay. There are no specifications for subjects based on age, race, sex or any other demographic. However, demographic information will be collected for each subject.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
PPA and NPA | In 7 days after specimen collection
  PPA and NPA between the VitaSIRO solo™ SARS-CoV-2/Flu/RSV and Cepheid Xpert® Xpress CoV-2/Flu/RSV plus assay

SECONDARY OUTCOMES:
Comparison to SOC testing | In 7 Days after specimen collection
  Evaluation of Diagnostic Performance Metrics for the VitaSIRO solo™ SARS-CoV-2/Flu/RSV Assay: Sensitivity, Specificity, PPV, and NPV Using Nasal and Nasopharyngeal Swabs Compared to Standard-of-Care Diagnostics

CONTACTS AND LOCATIONS:
Locations (1):
- Credo Diagnostics Biomedical Pte Ltd. Taiwan Branch, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truwit JD, Fleming K, Nanchal RS. Empowering Respiratory Therapists to Restrict Nebulized 3% Saline and N-Acetylcysteine During Mechanical Ventilation. Respir Care. 2025 Aug;70(8):937-945. doi: 10.1089/respcare.12586. Epub 2025 Feb 24. PMID 40028879